CLINICAL TRIAL: NCT05288296
Title: The Effect of Dynamic Taping to Improve the Landing Strategy in Athletes.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202002434B0
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-03

CONDITIONS: Landing Error Scoring System (LESS)
Keywords: Dynamic taping; Landing Error Scoring System (LESS); ACL injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Athletes in Taiwan (Experimental): In the first year, we would recruit senior high school soccer athletes (n=30) to observe the difference with/without dynamic taping on landing error scoring system under fatigue status. (2x2 cross-over study)
  In the second year, we would recruit junior/senior high school and college athlete (n=900) to establish a native model of single-leg and double-leg LESS, then in advanced, confirm the ability to predict ACL injuries.
  In the third year, we will focus on high-risk subjects evaluated by LESS and athlete with ACL reconstruction (n=60) to observe the supportive effect of dynamic taping. (2x2 cross-over study)
  Interventions: Device: dynamic taping

INTERVENTIONS:
Device: dynamic taping — 1. The intervention of dynamic tape can improve the LESS, which also means that we may reduce the probability of ACL injury through the intervention of dynamic tape.
  2. By establish a native model of single-leg and double-leg LESS can predict the occurrence of ACL injury early and further prevent it.

SUMMARY:
This study will be conducted in three years: In the first year, we would recruit male and female high school soccer athletes to observe the effect of dynamic taping on landing error scoring system under fatigue status. In the second year, we would recruit junior high school, high school and college athlete to establish a native model of single-leg and double-leg LESS, then in advanced, confirm the ability to predict ACL injuries. In the third year, we will focus on high-risk subjects evaluated by LESS and athlete with ACL reconstruction to observe the supportive effect of dynamic taping.

DETAILED DESCRIPTION:
ACL injuries occur most frequently in sports involving pivoting sudden deceleration. In Taiwan, it was estimated that at least 1,000 cases of patients require ACL reconstruction annually. Despite the improving of surgical technique, there is only 65% patients who received the ACL reconstruction return to their pre-injury level of sport. Therefore, to prevent ACL injuries in athletes is critical.

According to previous studies, the Landing Error Scoring System (LESS) is a clinical assessment tool to do field evaluation. We could predict the possibility of ACL injuries by the change of biomechanics. However, there are still many factors affecting the LESS, such as fatigue, single or double leg landing, age, sex and specific sport...etc., and comprehensive studies are absent.

Dynamic taping is a newly developing technique with better elasticity and extensibility. Studies showed that dynamic taping improve the biomechanics of knee joint. Hence, we can adjust the faulty movement as soon as possible to prevent the occurrence of ACL injuries.

This study will be conducted in three years: In the first year, we would recruit male and female high school soccer athletes to observe the effect of dynamic taping on landing error scoring system under fatigue status. In the second year, we would recruit junior high school, high school and college athlete to establish a native model of single-leg and double-leg LESS, then in advanced, confirm the ability to predict ACL injuries. In the third year, we will focus on high-risk subjects evaluated by LESS and athlete with ACL reconstruction to observe the supportive effect of dynamic taping.

ELIGIBILITY:
Inclusion Criteria:

* 1st Year: senior high school soccer athletes
* 2nd Year: junior/senior high school and college athlete
* 3dr Year: high-risk subjects evaluated by LESS and athlete with ACL reconstruction

Exclusion Criteria:

* Those who are unable to exercise due to acute joint, muscle or nerve injury in the lower extremities
* Lower extremity surgery within 1 year
* Head trauma within 6 months
* Those with vestibular injury within 6 months
* Allergic to Dynamic tape
* Pregnant
* Visual coordination impairment

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 990 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Landing Error Scoring System (LESS) Score | 1st Year
  Recruit senior high school soccer athletes (n=30) to observe the difference with/without dynamic taping on landing error scoring system under fatigue status. The Landing Error Scoring System (LESS) with double-leg consists of 17 items, total score is 0-19 points, whereas the single-leg consists of 14 items and total score is 0-16 points. Higher scores mean a worse outcome.
Landing Error Scoring System (LESS) Score | 2nd Year
  Recruit junior/senior high school and college athlete (n=900) to establish a native model of single-leg and double-leg LESS. The Landing Error Scoring System (LESS) with double-leg consists of 17 items, total score is 0-19 points, whereas the single-leg consists of 14 items and total score is 0-16 points. Higher scores mean a worse outcome.
Landing Error Scoring System (LESS) Score | 3rd Year
  Recruit high-risk subjects evaluated by LESS and athlete with ACL reconstruction (n=60) to observe the supportive effect of dynamic taping. The Landing Error Scoring System (LESS) with double-leg consists of 17 items, total score is 0-19 points, whereas the single-leg consists of 14 items and total score is 0-16 points. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: CHIH-KUAN WU, MD, Principal Investigator — Taoyuan Chang Gung Memorial Hospital, Taoyuan, Taiwan
Locations (1):
- Taoyuan Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No